CLINICAL TRIAL: NCT06602245
Title: Multicenter Observational Prospective Open Pilot Study of Changes in the Total Clearance of Antibacterial Agents During Hemoperfusion Using Efferon LPS in Patients With Sepsis
Brief Title: Clearance of Antibacterial Agents During Hemoperfusion in Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-lps-2024-01
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; Antibiotic clearance; Hemoperfusion; Extracorporeal therapy; Lipopolysaccharide sorption
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemoperfusion and antibiotic tratment groups: The trial will be conducted in one group of patients. Patients who are undergoing antibiotic therapy and hemoperfusion will be included in the study.
  Efferon LPS, a medical device, which is a single-use cartridge filled with a polymeric adsorbent that selectively adsorbs endotoxin via surface-immobilized ligand and excessive cytokines via its intrinsic porosity. All patients included undergo a single extracorporeal blood purification for 4-12 hours in the form of isolated hemoperfusion using the Efferon LPS device in combination with antibiotic therapy.
  The hemoperfusion must be started no later than 30 minutes after the end of the antibacterial drug administration, otherwise the patient will be excluded from the study.
  Antibacterial drugs are administered by infusion according to the instructions for use:
  * Meropenem within 30 minutes
  * Vancomycin within 60 minutes
  * Linezolid within 60 minutes.

SUMMARY:
One of the significants health problems in the world is sepsis, with the number of cases reaching 20-30 million per year, according to the WHO. Numerous studies have shown that the use of extracorporeal methods improves outcomes in patients with septic shock. Safety parameters are particularly important in deciding whether to initiate such therapy in a patient. To date, numerous post-marketing observations and data from the published literature have shown no serious adverse hemoperfusion events, with the exception of occasional thrombocytopenia. However, the potential removal of life-saving drugs, such as antibiotics, by hemoperfusion in patients with sepsis remains poorly understood and requires special attention.

The main objective of this study is to evaluate the incremental increase in total clearance of antibacterial drugs during haemoperfusion using the Efferon LPS device in patients with sepsis.

DETAILED DESCRIPTION:
Sepsis is a major public health problem worldwide, with 20-30 million cases per year according to the WHO. Lipopolysaccharide adsorption is used for the rapid resolution of the severe symptom complex associated with sepsis and septic shock. To date, numerous post-approval observations and data from the published literature have shown no serious adverse hemoperfusion events, except for occasional thrombocytopenia. At the same time, it is very important in the treatment of sepsis to start antibacterial drugs as early as possible, and the effect of lipopolysaccharide and cytokine adsorption on the clearance of antibacterial drugs remains poorly understood.

Little is known about the effects of modern sorption devices on the pharmacokinetics of antimicrobial drugs. The results obtained in animals and reports of single patient studies, as well as the results of in vitro studies, cannot be extrapolated to the general population of sepsis patients receiving hemoperfusion for the underlying disease. The observations need to be confirmed in clinical trials in patients with sepsis and septic shock in order to develop appropriate recommendations for dose adjustment of the antibacterial drugs used.

The present study in patients with sepsis and/or septic shock is designed to determine the effect of lipopolysaccharide adsorption using the Efferon LPS device on the pharmacokinetics of several antimicrobial agents (meropenem, vancomycin and linezolid).

ELIGIBILITY:
Inclusion Criteria:

* Patient weight greater than 40 kg.
* Diagnosis of sepsis and/or septic shock according to CEPSIS-3 criteria (2016), presumed (at time of enrolment) to be of Gram-negative aetiology, requiring, in the opinion of the investigator, isolated lipopolysaccharide hemoperfusion.

Exclusion Criteria:

* Failure to obtain informed consent from the patient, family member or legal representative.
* Any patient condition requiring other methods of renal replacement therapy (e.g. hemodialysis, hemofiltration, hemodiafiltration).
* Pregnancy, breastfeeding period.
* General contraindications to extracorporeal treatments.
* Any other condition that, in the opinion of the investigator, would prevent the patient from being a suitable candidate for inclusion in the study (e.g. terminal chronic disease).
* Development of an adverse event, including a serious adverse event; individual intolerance to the investigational product, hypersensitivity to the components of the product due to which further participation in the study is not possible.
* Continued participation in the study is not, in the opinion of the investigator, in the best interests of the patient's health.
* The patient, in the opinion of the investigator, fails to comply with the requirements of the study procedures.
* The presence of protocol deviations that, in the opinion of the Sponsor and the investigator, require withdrawal of the participant from the study.
* A positive pregnancy test result at any time during the study.
* Use of any other methods of renal replacement therapy and extracorporeal hemocorrection during isolated hemoperfusion with the Efferon LPS device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The expected number of study subjects is 30 adult patients with sepsis and/or septic shock (presumably of Gramnegative aetiology and any localisation).
  It is planned to recruit :
  * 10 patients receiving meropenem
  * 10 patients receiving vancomycin
  * 10 patients receiving linezolid. Patients may receive more than one of these antibiotics at the same time, in which case they will be included in several subpopulations of the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Adsorption clearance of antibacterial drugs by the Efferon LPS | During hemoperfusion with Efferon LPS
  Adsorption сlearance of antibacterial drugs by the Efferon LPS device, mL/min

SECONDARY OUTCOMES:
Total clearance of antibacterial drugs during haemoperfusion with the Efferon LPS | During hemoperfusion with Efferon LPS
  Total clearance of antibacterial drugs (adsorption clearance + patient system clearance), mL/min
Contribution of adsorption clearance to the total clearance of antibacterial drugs | During hemoperfusion with Efferon LPS
  Efferon LPS device adsorption clearance relative to total clearance, %

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Rey, PhD, MD, Principal Investigator — N. V. Sklifosovsky Moscow Research Institute of Emergency, Moscow, Russia
Locations (4):
- Russia (4):
  - N. V. Sklifosovsky Moscow Research Institute of Emergency, Moscow
  - N.I. Pirogov City Clinical Hospital No. 1, Moscow
  - Nizhny Novgorod Regional Clinical Hospital named after N.A. Semashko, Nizhny Novgorod
  - Perm regional clinical hospital, Perm